CLINICAL TRIAL: NCT02731235
Title: High-intensity Training in Patients With Lacunar Stroke (HITPALS)
Brief Title: The Effect of Aerobic Exercise in Patients With Lacunar Stroke
Acronym: HITPALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: University of Copenhagen (Other); Association of Danish Physiotherapists (Other)
Responsible Party: Principal Investigator, Christina Kruuse, Associate professor, consultant neurologist, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-15012371
Record Dates: First submitted 2016-01-22; First posted 2016-04-07 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Stroke, Lacunar
Keywords: Stroke; stroke, acute; Cerebral small vessel disease
MeSH Terms: conditions — Stroke, Lacunar; Stroke; Cerebral Small Vessel Diseases | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Prophylactic stroke medication and recommendations for lifestyle changes
  Interventions: Drug: prophylactic stroke medication; Behavioral: Recommendations for lifestyle changes
- Exercise (Active Comparator): Prophylactic stroke medication and recommendations for lifestyle changes AND high-intensity training at home, 5 days a week in 12 weeks
  Interventions: Other: High-intensity training; Drug: prophylactic stroke medication; Behavioral: Recommendations for lifestyle changes

INTERVENTIONS:
Other: High-intensity training — high intensity training 5 days a week for 12 weeks
  Arms: Exercise
Drug: prophylactic stroke medication — Usual care medication for stroke prophylaxis
Behavioral: Recommendations for lifestyle changes — Advise on diet, alcohol, smoking and exercise

SUMMARY:
In a randomized-controlled study the effect of high-intensity training, 5 days a week at home for 12 weeks is tested in patients with lacunar stroke.

DETAILED DESCRIPTION:
Little is known about effect of exercise for patients with lacunar stroke, no studies have investigated the feasibility or effect of aerobic exercise in this subgroup of stroke. The patients have few and temporary symptoms and are therefore early discharged from the hospital. After an cerebral infarct the patients have increased risk of recurrent stroke and they are at risk of developing cognitive deficits or vascular dementia over time. Researchers want to investigate if high-intensity training at home in the acute phase has an effect on aerobic fitness, endothelial response and health profile in this potential fragile group of patients. We hope to increase the patients´ physical and mental function, and thereby prevent a recurrent stroke and slow the progression of vascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* lacunar stroke verified by clinical examination and CT- or MRI-scans
* able to speak and read Danish

Exclusion Criteria:

* previous large artery stroke,
* symptoms or co-morbidities in the musculoskeletal system, which hinder bicycling,
* dyspnoea caused by heart or pulmonary disease,
* aphasia or dementia which hinder completion of the Talk Test.

Amendment 1 (version 4.0, June 2016) has been modified to allow an extended inclusion period from 0-21 days (previously 0-7 days).

Also, to allow inclusion of patients with recurrent lacunar stroke, with clinical symptoms and a corresponding ischemic lesion on MRI.

Amendment 2 (version 5.0, June 2017) has allowed inclusion from two other stroke units in the Capital Region of Copenhagen due to low recruitment rate. The article describes protocol version 5.0 from June 6th. 2017

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Difference in the 'Graded Cycling Test with Talk Test' | at baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  Sub-maximal exercise test on a stationary bicycle

SECONDARY OUTCOMES:
Endothelial response | at baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  measurement of endothelial response by Endopat2000
Physical Activity Scale (PAS) | at baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  A questionnaire that measures the level of self-reported physical activity
Short time activity measurements | at baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  Accelerometer (Axivity) to short time registration of physical activity (24 hours in an 8 day period (after inclusion, before 3 months visit, before 12 month visit)
The WHO-five Well-being Index (WHO-5) | at baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  A questionnaire that measures current mental well-being
Montreal Cognitive Assessment (MOCA) | at baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  A cognitive screening test for detection of mild cognitive impairments
Major Depression Inventory (MDI) | at baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  A self-report mood questionnaire
Multidimensional Fatigue Inventory (MFI-20) | at baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  A 20-item self-report instrument designed to measure fatigue.
Ull-Meter | At baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  An instrument which measures the individual stress reaction - it presents an objective number for the body and mind's state of stress.
Blood samples | at baseline, 3 (primary analysis), 6 and 12 months after baseline testing
  Blood samples to determine cardiovascular risk factors
Magnetic resonance Imaging (MRI) | 12 months after baseline testing
  Detection of new infarcts or white matter lesions

OTHER OUTCOMES:
Cardio-vascular event or death | 5 years
  Follow-up 5 years from inclusion on cardiovascular events or death

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kruuse, MD, DMSc, Principal Investigator — Herlev Hospital, Dept Neurology
Locations (1):
- Herlev Hospital, Dept Neurology, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251
- [Derived] Steen Krawcyk R, Vinther A, Petersen NC, Faber J, Iversen HK, Christensen T, Lambertsen KL, Rehman S, Klausen TW, Rostrup E, Kruuse C. Effect of Home-Based High-Intensity Interval Training in Patients With Lacunar Stroke: A Randomized Controlled Trial. Front Neurol. 2019 Jun 28;10:664. doi: 10.3389/fneur.2019.00664. eCollection 2019. PMID 31316451